CLINICAL TRIAL: NCT01650246
Title: A Long-Term Open-Label Extension Study for Subjects Completing a Phase 3 Efficacy and Safety Study of Lesinurad Monotherapy in Subjects With Gout
Brief Title: Open-Label Lesinurad Monotherapy Extension Study in Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDEA594-305
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lesinurad 400 mg (Experimental)
  Interventions: Drug: lesinurad

INTERVENTIONS:
Drug: lesinurad — Tablets, 400 mg QD

SUMMARY:
This study will assess the serum uric acid lowering effects and safety of lesinurad over a long-term timeframe.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, uncontrolled, extension study to assess the long-term efficacy and safety of lesinurad monotherapy in subjects who completed the double-blind treatment period in Study RDEA594-303.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures and the risks involved and is willing to provide written informed consent before the first study related activity.
* Subject completed the double-blind treatment period in Study RDEA594-303 and was actively receiving and tolerating study medication (lesinurad or placebo) at Month 6 visit.
* Subject is willing to adhere to the visit/protocol schedules.
* Subject is male or female; female subjects of childbearing potential must agree to use an effective non-hormonal method of birth control during the study and for at least 14 days after the last dose of study medication.

Exclusion Criteria:

* Subject has any other medical or psychological condition, which in the opinion of the Investigator and/or the Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or to complete the study.
* Subject has a past medical history of urolithiasis, nephrolithiasis, or kidney stone diathesis.
* Subject developed kidney stones during Study RDEA594-303

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Director — Ardea Biosciences, Inc.
Locations (72):
- United States (54):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Peoria, Arizona
  - Tempe, Arizona
  - Carmichael, California
  - Covina, California
  - Huntington Park, California
  - Irvine, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - Trumbill, Connecticut
  - Boynton Beach, Florida
  - Miami, Florida
  - Plant City, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Newnan, Georgia
  - Honolulu, Hawaii
  - Meridian, Indiana
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Metairie, Louisiana
  - Traverse City, Michigan
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - New Windsor, New York
  - New York, New York
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Perrysburg, Ohio
  - Jenkintown, Pennsylvania
  - Landsdale, Pennsylvania
  - Sellersville, Pennsylvania
  - Myrtle Beach, South Carolina
  - Spartanburg, South Carolina
  - Brentwood, Tennessee
  - Spring Hill, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Bountiful, Utah
  - West Layton, Utah
  - Chesapeake, Virginia
  - Richmond, Virginia
  - Suffold, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
- Australia (2):
  - Herston, Queensland
  - Hobart, Tasmania
- Belgium (4):
  - Genk
  - Gozée
  - Kortrijk
  - Yvoir
- Canada (3):
  - Toronto, Ontario
  - Québec, Quebec
  - Rimouski, Quebec
- Germany (2):
  - Dresden
  - Leipzig
- New Zealand (2):
  - Grafton, Auckland
  - Tauranga
- South Africa (5):
  - Silverglen, Durban
  - Muckleneuk, Pretoria
  - Rondebosch
  - Stellenbosch
  - Thabazimbi

RESULTS

PARTICIPANT FLOW:
Groups:
- Lesinurad 400 mg: lesinurad 400 mg once daily (qd)
Period: Overall Study
Arm/Group | Lesinurad 400 mg
Started | 143
Completed | 0
Not Completed | 143
Not completed — Adverse Event | 23
Not completed — Protocol Violation | 5
Not completed — Sponsor terminated study | 53
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 26
Not completed — Death | 1
Not completed — Lack of Efficacy | 30

BASELINE CHARACTERISTICS:
Arm/Group | Lesinurad 400 mg
Number analyzed (Participants) | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.0)
Age, Customized [Number; unit: Participants] — <65 Years, >=65 Years
  Participants
    <65 Years | 111
    >=65 Years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 132
Region of Enrollment [Number; unit: Participants]
  Australia | 2
  Belgium | 9
  Canada | 6
  Germany | 6
  New Zealand | 3
  South Africa | 16
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Serum Urate (sUA) Level That is < 6.0 mg/dL
Time Frame: Month 1
Population: Safety Population
Measure: Number; unit: Subjects
Arm/Group | Lesinurad 400 mg
Number analyzed (Participants) | 143
Subjects | 68

2. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Time Frame: Up to approximately 2 years
Population: Safety Population
Measure: Number; unit: TEAEs
Arm/Group | Lesinurad 400 mg
Number analyzed (Participants) | 143
TEAEs | 105

ADVERSE EVENTS:
Arm/Group | Lesinurad 400 mg
Serious Adverse Events (participants affected / at risk) | 15/143
Other Adverse Events (participants affected / at risk) | 73/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 400 mg (N=143)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrioventricular clock complete (Cardiac disorders) | 1 (1)
Coronary Artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 400 mg (N=143)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (7)
Fatigue (General disorders) | 4 (4)
Pyrexia (General disorders) | 3 (3)
Bronchitis (Infections and infestations) | 5 (5)
Gastroenteritis (Infections and infestations) | 7 (8)
Influenza (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 14 (15)
Urinary tract infection (Infections and infestations) | 7 (8)
Blood creatine phosphokinase increased (Investigations) | 4 (4)
Blood creatinine increased (Investigations) | 16 (20)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 6 (8)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Renal impairment (Renal and urinary disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypertension (Vascular disorders) | 10 (10)
Nasopharyngitis (Infections and infestations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.